CLINICAL TRIAL: NCT00833924
Title: Evaluation of the Safety and Effectiveness of the Zenith(R) Low Profile AAA Endovascular Graft
Brief Title: Zenith(R) Low Profile AAA Endovascular Graft Clinical Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cook Group Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 08-013; 370016
Expanded Access: NCT02557659 (No longer available)
Record Dates: First submitted 2009-01-30; First posted 2009-02-02 (Estimated); Results first posted 2016-01-29 (Estimated); Last update posted 2018-04-04 (Actual); Status verified 2018-03

CONDITIONS: Abdominal Aortic Aneurysms; Iliac Aneurysms; Aorto-iliac Aneurysms
Keywords: Low Profile; Abdominal Aortic Aneurysms; Endovascular
MeSH Terms: conditions — Aortic Aneurysm, Abdominal; Iliac Aneurysm

ARMS (1):
- 1 (Other): Treatment with Endovascular Graft
  Interventions: Device: Zenith(R) Low Profile AAA Endovascular Graft

INTERVENTIONS:
Device: Zenith(R) Low Profile AAA Endovascular Graft — The Zenith(R) Low Profile AAA Endovascular Graft and ancillary components are indicated for the endovascular treatment of patients with abdominal aortic, aorto-iliac, or iliac aneurysms having morphology suitable for endovascular repair.

SUMMARY:
The Zenith® Low Profile AAA Endovascular Graft Clinical Study is a clinical trial approved by US FDA to study the safety and effectiveness of the Zenith® Low Profile AAA Endovascular Graft to treat abdominal aortic, aorto-iliac, and iliac aneurysms.

ELIGIBILITY:
Inclusion Criteria:

* Abdominal aortic, aortoiliac, and iliac aneurysms of appropriate size
* Vessels suitable for endovascular access and aneurysm repair

Exclusion Criteria:

* Less than 18 years of age
* Inability or refusal to give informed consent
* Disease considerations that would compromise patient safety or study outcomes
* Unsuitable arterial anatomy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2008-05; Primary Completion 2011-10 (Actual); Study Completion 2016-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ronald Fairman, MD, Principal Investigator — University of Pennsylvania
Locations (27):
- United States (23):
  - University of California, San Francisco, Div. Vascular Surgery and San Francisco VAMC, San Francisco, California
  - Stanford University Medical Center, Stanford, California
  - Yale New Haven School of Med., Dept. of Vascular Surgery, New Haven, Connecticut
  - University of Florida, Vascular Surgery, Gainesville, Florida
  - Massachusetts General Hospital, Boston, Massachusetts
  - University of Michigan Hospital, Ann Arbor, Michigan
  - Spectrum Health Butterworth, Grand Rapids, Michigan
  - William Beaumont Hospital, Royal Oak, Michigan
  - Mayo Clinic, Rochester, Minnesota
  - Barnes-Jewish Hospital, St Louis, Missouri
  - Mercy Hospital, St Louis, Missouri
  - Morristown Memorial Hospital, Morristown, New Jersey
  - New York University Hospital, New York, New York
  - New York Presbyterian Hospital - Cornell, New York, New York
  - University of Rochester, Strong Memorial Hospital, Rochester, New York
  - University of North Carolina, Chapel Hill, North Carolina
  - Cleveland Clinic, Cleveland, Ohio
  - Ohio Health Research Institute, Columbus, Ohio
  - Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
  - Allegheny General Hospital, Pittsburgh, Pennsylvania
  - Fairfax Inova Hospital, Falls Church, Virginia
  - Harborview Medical Center, Seattle, Washington
  - St. Luke's Medical Center, Milwaukee, Wisconsin
- Queen Mary Hospital, Hong Kong, China
- St. Franziskus Hospital, Münster, Germany
- CELT Hospital, Moscow, Russia
- Malmo University Hospital, Malmo, Sweden

RESULTS

PARTICIPANT FLOW:
Groups:
- Zenith® Low Profile AAA Endovascular Graft: The Zenith® Low Profile AAA Endovascular Graft and ancillary components are indicated for the endovascular treatment of patients with abdominal aortic, aorto-iliac, or iliac aneurysms having morphology suitable for endovascular repair.
Period: Overall Study
Arm/Group | Zenith® Low Profile AAA Endovascular Graft
Started | 120
30-day | 120
12-month | 113
Completed | 11
Not Completed | 109
Not completed — Death | 21
Not completed — Conversion | 2
Not completed — Lost to Follow-up | 2
Not completed — Withdrawal by Subject | 13
Not completed — In study follow-up | 71

BASELINE CHARACTERISTICS:
Arm/Group | Zenith® Low Profile AAA Endovascular Graft
Number analyzed (Participants) | 120
Age, Continuous [Mean (Standard Deviation); unit: years] | 71.8 (8.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16
  Male | 104

OUTCOME MEASURES:

1. Primary Outcome: Patients With Major Adverse Events (MAE)
Description: MAE is defined as any occurrence of all-cause death, Q-wave myocardial infarction (MI), renal failure requiring dialysis, paralysis, stroke, bowel ischemia, or re-intubation.
Time Frame: 30-day
Population: 1 patient experienced a re-intubation, which was adjudicated by the CEC as not related to AAA repair (related to a pre-existing condition).
Measure: Number; unit: participants
Arm/Group | Zenith® Low Profile AAA Endovascular Graft
Number analyzed (Participants) | 120
participants | 1
Statistical Analysis 1: Comparison: Zenith® Low Profile AAA Endovascular Graft; Null hypothesis: The 30-day Freedom from MAE for patients treated with the Zenith® Low Profile AAA Endovascular Graft does not meet the performance goal (88%); Test type: Superiority or Other; p < 0.01, Exact binomial test; Rate of 30-day freedom from MAE = 99.2, 95% CI 2-sided [95.4 to 100]

2. Primary Outcome: Patients With Device Failures
Description: Device success at 12-month is defined as:
  Technical Success (successful access of the aneurysm site, deployment of the graft in the intended location, and patency of the graft at the time of deployment completion intra-operatively), and freedom from the following at 12 months: Type I or type III endoleaks requiring re-intervention, Aneurysm rupture or conversion to open surgical repair, and Aneurysm enlargement greater than 0.5 cm.
Time Frame: 12-month
Population: There were 5 patients died, and 2 patients withdrew.
Measure: Number; unit: participants
Arm/Group | Zenith® Low Profile AAA Endovascular Graft
Number analyzed (Participants) | 113
participants
  Converted to open surgical repair | 1
  Aneurysm expansion > 5 mm | 2
Statistical Analysis 1: Comparison: Zenith® Low Profile AAA Endovascular Graft; Null hypothesis: The 12-month device success for patients treated with the Zenith® Low Profile AAA Endovascular Graft does not meet the performance goal (84%); Test type: Superiority or Other; p < 0.01, Exact binomial test; 12-month Device Success Rate = 97.3, 95% CI 2-sided [92.4 to 99.4]

ADVERSE EVENTS:
Time Frame: 365 days
Arm/Group | Zenith® Low Profile AAA Endovascular Graft
Serious Adverse Events (participants affected / at risk) | 63/120
Other Adverse Events (participants affected / at risk) | 8/120
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Zenith® Low Profile AAA Endovascular Graft (N=120)
Anemia (Blood and lymphatic system disorders) | 1 (1)
Hypoglycemia (Blood and lymphatic system disorders) | 1 (1)
Iron deficiency anemia requiring transfusion (Blood and lymphatic system disorders) | 1 (1)
Leukocytosis with fever (Blood and lymphatic system disorders) | 1 (1)
Low hemoglobin (6.9) transfused 2 units packed red blood cells (PRBC) (Blood and lymphatic system disorders) | 1 (1)
Arrhythmia requiring intervention or new treatment (Cardiac disorders) | 5 (5)
Bradycardia (Cardiac disorders) | 1 (1)
Cardiac event involving arrest, resuscitation, or balloon pump (Cardiac disorders) | 1 (1)
Cardiac ischemia requiring intervention (Cardiac disorders) | 1 (1)
Chest discomfort (Cardiac disorders) | 1 (1)
Chest pain requiring hospital admission and cardiac catheterization (Cardiac disorders) | 1 (1)
Congestive Heart Failure (Cardiac disorders) | 3 (3)
Episode of supraventricular tachycardia (Cardiac disorders) | 1 (1)
Hypertension (Cardiac disorders) | 1 (1)
Hypotension (Cardiac disorders) | 1 (2)
New onset sinus tachycardia (Cardiac disorders) | 1 (1)
Non-cardiac chest pain (Cardiac disorders) | 1 (1)
Syncope due to symptomatic bradycardia (Cardiac disorders) | 1 (1)
Uncontrolled hypertension (Cardiac disorders) | 1 (1)
Upgrade of an implantable cardioverter (ICD) to a BIV ICD as well as implantation of a new ICD lead (Cardiac disorders) | 1 (1) — BIV stands for biventricular
Cataract removal (left eye) (Eye disorders) | 1 (1)
Abdominal incisional hernia repair (Gastrointestinal disorders) | 1 (1)
Abdominal pain, distention, hematemesis (Gastrointestinal disorders) | 1 (1)
Abdominal wall seroma (Gastrointestinal disorders) | 1 (1)
Abscess (Gastrointestinal disorders) | 1 (1)
Acute diverticulitis in the descending colon (Gastrointestinal disorders) | 1 (1)
Aspiration with paraesophageal hernia (Gastrointestinal disorders) | 1 (1)
Bowel resection (Gastrointestinal disorders) | 1 (1)
Cellulitis to the abdominal wall (Gastrointestinal disorders) | 1 (1)
Gastritis with epigastric pain (Gastrointestinal disorders) | 1 (1)
Gastrointestinal bleeding requiring treatment (Gastrointestinal disorders) | 2 (2)
Gastrointestinal infection requiring treatment (Gastrointestinal disorders) | 1 (1)
Possible colonic ileus (Gastrointestinal disorders) | 1 (1)
Right inguinal hernia (Gastrointestinal disorders) | 1 (1)
Cellulitis (Infections and infestations) | 1 (1)
Sepsis (Infections and infestations) | 3 (3)
Complication requiring return to operating room (OR) (Injury, poisoning and procedural complications) | 1 (1)
Penile/bilateral groin ecchymosis/swelling (Injury, poisoning and procedural complications) | 1 (1)
Perineal wound discharge after resection of rectum (Injury, poisoning and procedural complications) | 1 (1)
Fall resulting in rib fracture and closed fracture of acetabulum (Injury, poisoning and procedural complications) | 1 (1)
Seroma requiring treatment (Injury, poisoning and procedural complications) | 1 (1)
Wound infection requiring antibiotic treatment (Injury, poisoning and procedural complications) | 4 (4)
Found to have diabetes (Metabolism and nutrition disorders) | 1 (1)
New diagnosis of hyperthyroidism (Metabolism and nutrition disorders) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Left hip pain due to degeneration of hip joint (Musculoskeletal and connective tissue disorders) | 1 (1)
Left knee degenerative joint disease (Musculoskeletal and connective tissue disorders) | 2 (2)
Pain left calf on exertion (Musculoskeletal and connective tissue disorders) | 1 (1)
Lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Prostate cancer diagnosed by biopsy (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
T1 grade 3 urothelial carcinoma of the bladder (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Altered mental status (Nervous system disorders) | 2 (2)
Encephalopathy (Nervous system disorders) | 1 (1)
Left partial third nerve palsy. Diplopia. (Nervous system disorders) | 1 (1)
Paresthesias associated with limb ischemia (Nervous system disorders) | 1 (1)
Stroke (Nervous system disorders) | 1 (1)
Acute renal failure (Renal and urinary disorders) | 1 (1)
Hematuria (Renal and urinary disorders) | 1 (1)
Kidney stone (Renal and urinary disorders) | 1 (1)
Left renal atrophy and scarring (Renal and urinary disorders) | 1 (1)
Penile cellulitis (Renal and urinary disorders) | 1 (1)
Renal failure requiring dialysis (Renal and urinary disorders) | 1 (1)
Retention of urine (Renal and urinary disorders) | 1 (1)
Right nephrectomy (Renal and urinary disorders) | 1 (1)
Serum creatinine rise > 30% above baseline resulting in a persistent value > 2.0 mg/dl (Renal and urinary disorders) | 2 (2)
Urethral stricture (Renal and urinary disorders) | 1 (1)
Urinary retention (Renal and urinary disorders) | 2 (2)
Urinary tract infection (UTI) requiring antibiotic treatment (Renal and urinary disorders) | 6 (7)
Epididymitis and fever (Reproductive system and breast disorders) | 1 (1)
Right hydrocele (Reproductive system and breast disorders) | 1 (1)
Acute chronic obstructive pulmonary disease (COPD) exacerbation (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Exacerbation of asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hypoxemia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Increased dyspnea leading to new diagnosis of sleep apnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
New 7.7 cm right upper lung zone mass concerning for neoplasm (Respiratory, thoracic and mediastinal disorders) | 1 (1)
New diagnosis of sleep apnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Persistent left lung atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pleural effusion requiring treatment (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pnuemonia requiring antibiotics (Respiratory, thoracic and mediastinal disorders) | 5 (5)
Pulmonary event requiring tracheostomy or chest tube (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Re-intubation (Respiratory, thoracic and mediastinal disorders) | 1 (3)
Shortness of breath with right swollen extremity (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Percutaneous endoscopic gastrostomy (PEG) placement (Surgical and medical procedures) | 1 (1)
Arterial thrombosis in graft (Vascular disorders) | 9 (11)
Arterial thrombosis in native artery (Vascular disorders) | 3 (3)
Bilateral popliteal aneurysms/left side thrombosed (Vascular disorders) | 1 (1)
Claudication (Vascular disorders) | 1 (1)
Clotted left superficial femoral artery (LSFA) to post-tibial bypass graft (Vascular disorders) | 1 (1)
Embolization resulting in tissue loss or requiring intervention (Vascular disorders) | 5 (7)
Hematoma (Vascular disorders) | 2 (2)
Hematoma requiring surgical repair (Vascular disorders) | 1 (2)
Left lower extremity aneurysm (Vascular disorders) | 1 (1)
Low systolic blood pressure: 70 recorded on 10/14/09 (Vascular disorders) | 1 (1)
Non-occlusive graft thrombus (Vascular disorders) | 9 (10)
Patient became hypotensive upon anesthesia induction - sustained (Vascular disorders) | 1 (1)
Post-procedure transfusion (Vascular disorders) | 6 (6)
Right leg pulselessness (Vascular disorders) | 1 (1)
Vascular injury (Vascular disorders) | 3 (3)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Zenith® Low Profile AAA Endovascular Graft (N=120)
Post-procedure transfusion (Vascular disorders) | 8 (8)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days